CLINICAL TRIAL: NCT05286879
Title: Addressing Risk Through Community Treatment for Infectious Disease and Opioid Use Disorder Now (ACTION) Among Justice-involved Populations
Acronym: ACTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000029346; 1U01DA053039-01 (NIH)
Record Dates: First submitted 2022-02-25; First posted 2022-03-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Infectious Disease; Risk Reduction Behavior; Substance Use; Substance Abuse; Stimulant Use Disorder
Keywords: Justice involvement; HIV Prevention; Hepatitis C Prevention
MeSH Terms: conditions — Opioid-Related Disorders; Communicable Diseases; Risk Reduction Behavior; Substance-Related Disorders | interventions — Patient Navigation; Mobile Health Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigator (Other): Navigators will assist linking study participants to appropriate community service providers
  Interventions: Behavioral: Patient Navigator
- Mobile Health Unit (Other): Study participants will be linked to a MHU within their community
  Interventions: Behavioral: Mobile Health Unit

INTERVENTIONS:
Behavioral: Patient Navigator — Linkage to services for OUD/SUD treatment including MOUD, Hepatitis C virus (HCV) testing and treatment; those not living with HIV infection will be provided access to PrEP services, and those living with HIV will receive assistance with gaining initial or continued access to ART services during the 6-month post-release intervention period
  Arms: Patient Navigator
Behavioral: Mobile Health Unit — Participants will receive HIV PrEP/ HIV ART, MOUD, harm reduction services on the MHU and or assistance from a community health worker in linking to appropriate community-based OUD and other medical and behavioral health providers across the 6 month post-release intervention period
  Arms: Mobile Health Unit

SUMMARY:
This is a 5-year Hybrid Type 1 Effectiveness-Implementation Randomized Control Trial (RCT) that compares two models of linking and retaining individuals recently released from justice involvement to the continuum of community-based HIV prevention and treatment, HCV treatment, STI treatment, and opioid use disorder (OUD) prevention and treatment, medication for opioid use disorder (MOUD) service cascades of care.

DETAILED DESCRIPTION:
This 5-year Hybrid Type 1 Effectiveness-Implementation RCT trial compares two models of linking and retaining individuals recently released from justice involvement to the continuum of community-based HIV and OUD prevention and treatment (MOUD) service cascades of care. A significant innovation of this RCT is that it will be delivered within 4 communities where coalition infrastructures have been established as part of the Justice Community Opioid Innovation Network (JCOIN) studies, a National Institute on Drug Abuse (NIDA)-funded Cooperative Agreement initiative to mitigate the impact criminal justice (CJ)-involved individuals with OUD are having on local communities, and the investigators will be able to build on that existing infrastructure. Specifically, up to 960 CJ-involved individuals will be recruited across 2 CT (New London/Middlesex Counties and Windham/Tolland/New Haven/Hartford Counties) & 2 Texas (Dallas and Tarrant Counties) high risk communities. HIV status will be assessed via rapid testing at initial point of contact. Participants will be randomized to receive at post-release either: a) a Patient Navigator (PN) system for care, wherein navigators will assist linking study participants to appropriate community service providers (e.g., OUD/SUD treatment including MOUD, and HCV testing and treatment; those not living with HIV will be provided access to pre-exposure prophylaxis (PrEP) services, and those living with HIV will receive assistance with gaining initial or continued access to antiretroviral therapy (ART) services, or b) services delivered via a Mobile Health Unit (MHU) within the participants community where participants will receive PrEP/ART, MOUD, and harm reduction services on the MHU or assistance from a community health worker (CHW) in linking to appropriate community-based OUD and other medical and behavioral health providers. The interventions will last for 6 months post-release from custody. The focus of this study is the randomized controlled trial.

Study objectives:

Aim 1 (Intervention Effectiveness) Primary: To compare the effectiveness of PN vs. MHU service delivery on participant length of time to initiating post-release PrEP (prevention)/ART (treatment) medication within 6 months following release from justice involvement. Secondary outcomes will examine the continuum of PrEP and HIV care outcomes, including (but not limited to) the following additional HIV-related measures: viral suppression for people living with HIV (PLH), PrEP adherence, HIV risk behaviors; HCV Measures: HCV testing & linkage to treatment. Importantly, the investigators will also assess OUD and Substance Use Disorders (SUD)-related measures: OUD/SUD diagnoses, MOUD prescription receipt & retention, opioid & stimulant use, and overdose incidents. Other outcomes of interest include sexually transmitted infection (STI) incidence; and primary medical care appointments.

Aim 2 (Implementation): To evaluate Patient Navigation (PN ) and Mobile Health Unit (MHU) feasibility, acceptability, and costs. Primary implementation outcomes include feasibility (health care utilization impact among released individuals, contributions of interagency workgroup members on outcomes); acceptability (participant satisfaction, perceived usefulness); sustainment (continued utilization), and costs required to implement and sustain the approaches as well as to scale-up in additional communities. Additional outcomes will examine the broader impact on community health care including other health services accessed, expanded OUD services, and common barriers (e.g., stigma) to service access across the community provider spectrum. The investigators will also assess cost offsets and effectiveness of the service delivery models on the cascade outcomes. A Persons Who Inject Drugs (PWID) sub-study will focus on gaining insight into participant and social context (inner and outer) factors associated with the effectiveness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Living in one of our research areas
* Age 18 or older
* Able to provide written informed consent in English or Spanish
* Involvement with the criminal justice system within the last 6 months
* Living with HIV or being at risk of acquiring HIV and willing to learn about PrEP
* Willing to be tested for HIV (unless already confirmed via medical record)
* Having a history of opioid and/or stimulant use within 12 months prior to being in a controlled setting and/or in the last 6 months within the community
* Having a history of condomless sexual intercourse, STI diagnosis, and/or IDU within 6 months prior to being in a controlled setting and/or in the last 6 months within the community

Exclusion Criteria:

* Severe medical or psychiatric disability making participation unsafe
* Unable to provide consent
* Not remaining in the local area after release from custody
* Being released to inpatient care
* Potential risk to research staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to post-release initiation of ART medication | From the day of release/randomization to initiation of ART up to 6 months
  Time to post-release initiation of ART for persons living with HIV. Measured by self-reported initiation within 6-months. ART initiation will be measured as the date of self-reported initiation within the 6-month intervention period.
Time to post-release initiation of PrEP medication | From the day of release/randomization to initiation of PrEP up to 6 months
  Time to post-release initiation of PrEP for participants not living with HIV. Measured by self-reported initiation within 6-months. PrEP initiation will be measured as the date of self-reported initiation within the 6-month intervention period.

SECONDARY OUTCOMES:
Proportion of participants that initiate PrEP | From the day of release/randomization to initiation of PrEP up to 6 months
  The proportion of participants who initiate PrEP, of those who are not living with HIV, will be assessed via self-report and through confirmation with community provider
Proportion of participants prescribed PrEP at end of intervention. | 6 months
  Proportion of participants prescribed PrEP at end of intervention via self-report and through confirmation with community provider
PrEP adherence by self-report | 6 months
  For participants who initiate PrEP, adherence will be assessed by self-reported PrEP adherence via Visual Analog Scale (VAS)
Change in HIV status | Baseline and 12 months
  Change in HIV status for participants testing negative using rapid point of care (POC) via Orasure tests at baseline that have a follow-up reactive HIV point of care test
ART adherence by self-report | 6 months
  For PLH, adherence to ART treatment will be assessed by self-reported ART adherence via Visual Analog Scale (VAS)
HIV viral suppression | 6 months
  For PLH, HIV viral suppression, for those with HIV at time of randomization: the percent who maintain or achieve HIV viral load < 200 copies/mL at 6 months
HIV Risk behaviors | from baseline up to 6 months
  Changes in injection and sexual risk behaviors, a summary item from Dr. Springer's HIV Risk Behavior tool created for NIDA Small Business Technology Transfer (STTR) will be used to assess sharing of injection equipment and other drug and sexual risk behaviors
Type of opioids used | 6 months
  Type of opioids used (not as prescribed) will be assessed by the Texas Christian University Drug Screen 5.
Opioid abstinence | 6 months
  The percent of opioid-free months by self-report via the timeline followback (TLFB).
Substance use treatment participation | 6 months
  Substance use treatment participation will be collected via self-report. Treatments include detoxification, residential treatment, and medication treatments.
Type of substances used | 6 months
  Types of other substances used (e.g. stimulant, benzodiazepine, marijuana, synthetic cannabinoids, and alcohol) not as prescribed will be assessed self-reported via Texas Christian University Drug Screen 5
Substance use related overdoses at 6 months | 6 months
  Occurrence of non-fatal and fatal substance use related overdoses, through self-report, confirmation with medical providers, and mortality index data
Substance use related overdoses at 12 months | 12 months
  Occurrence of non-fatal and fatal substance use related overdoses, through self-report, confirmation with medical providers, and mortality index data

OTHER OUTCOMES:
PrEP adherence by dried blood spot (DBS) testing | 6 months
  For participants who initiate PrEP, adherence will be measured by DBS testing (Orasure, Inc.) and defined as a tenofovirdisoproxil diphosphate (TFV-DP) level >700 fmol/punch at 6 months, reflecting cumulative dosing over 6-8 weeks and consistent with 4 or more doses of PrEP per week.
PrEP adherence by urine sample analysis | 6 months
  For participants who initiate PrEP, adherence will be assessed by TFV-DP urine testing, which measures recent (past 48 hour) dosing (Orasure, Inc.)
PrEP adherence assessed by prescription refill data | up to 6 months
  For participants who initiate PrEP, the proportion who are adherent based on continuous PrEP prescription refill will be assessed by date of prescription refill and number of pills per refill, via pharmacy data.
Retention in HIV PrEP care | up to 6 months
  Retention in PrEP care defined as attending 2 or more visits in 6 months post-release will be assessed via self-report and through confirmation with community provider
ART adherence by DBS testing | 6 months
  For participants living with HIV (PLH), adherence to ART treatment measured via the dry blood spot for TFV-DP, level >700 fmol/punch at 6 months
ART adherence by urine sample analysis | 6 months
  For PLH, adherence to ART treatment measured via urine testing for TFV-DP based regimens.
ART adherence by prescription refill | up to 6 months
  For participants who are prescribed ART, the proportion who are adherent based on continuous ART prescription refill will be assessed by date of prescription refill and number of pills per refill, via pharmacy data.
Retention in HIV ART care | up to 6 months
  For PLH, retention in HIV ART care: defined as attending 2 or more visits in 6 months post-release will be assessed via selfreport and through confirmation with community provider
Hepatitis C incidence at baseline | at baseline
  The proportion who test positive on rapid POC Hepatitis C virus (HCV) test with confirmatory reflex HCV viral load at baseline
Hepatitis C incidence | 6 months
  The proportion who test positive on rapid POC HCV test with confirmatory HCV viral load at 6 months
Hepatitis C linkage | Day of release/randomization to appointment time up to 6 months
  Time to linked appointment for HCV treatment during the 6 month intervention will be assessed via self-report and through confirmation with community provider
Hepatitis C medication initiation via self-report | From baseline to reported treatment up to 6 months
  Time to HCV direct acting antiviral treatment (DAAs) during the 6 month will be assessed via self-report VAS
Hepatitis C medication initiation by prescription refill | up to 6 months
  HCV direct acting antiviral treatment (DAAs) during the 6 month will be assessed via prescription refill data
Hepatitis C medication initiation by confirmation from provider | up to 6 months
  Initiation of HCV direct acting antiviral treatment (DAAs) during the 6 month will be assessed via confirmation with community provider
Hepatitis C medication completion by self-report | 6 months
  The proportion of participants prescribed DAAs who complete treatment will be assessed via self-report at 6 months
Hepatitis C medication completion by prescription refill | 6 months
  The proportion of participants prescribed DAAs who complete treatment will be assessed via prescription refill data at 6 months
Hepatitis C medication completion by confirmation from provider | 6 months
  The proportion of participants prescribed DAAs, who complete treatment will be assessed via confirmation with community provider at 6 months
Hepatitis C sustained viral remission (SVR) | up to 6 months
  The proportion of participants who achieve SVR at week 12 upon completion of DAA prescription medication, assessed as undetectable HCV viral load.
Hepatitis C re-infection | 12 months
  The proportion of participants, of those that achieve HCV SVR, that are re-infected with HCV at 12 months, via reactive rapid HCV POC test result
Opioid use | 6 months
  Opioid use (not as prescribed) will be assessed by the proportion of monthly urine samples negative vs. positive/missing
Number of opioid use days | 6 months
  Number of days of opioid use, not as prescribed, will be assessed using the timeline follow back (TLFB) method
Linkage to medications for opioid use disorder (MOUD) via self-report | From day of release/randomization to appointment for MOUD up to 6 months
  Time to linked appointment for MOUD treatment during the 6 month intervention will be assessed via self-report
Linkage to medications for opioid use disorder (MOUD) via community provider | From day of release/randomization to appointment for MOUD up to 6 months
  Time to linked appointment for MOUD treatment during the 6 month intervention will be assessed via confirmation with community provider
MOUD retention by community provider | up to 6 months
  Retention on MOUD type and dose of MOUD via confirmation from community provider
MOUD retention by self-report | up to 6 months
  Retention on MOUD, using the Justice Community Opioid Innovation Network (JCOIN) instrument via self-reported type and dose of MOUD
Substance use | 6 months
  Use of other substances (e.g. stimulant, benzodiazepine, methylenedioxymethamphetamine, marijuana, and alcohol) not as prescribed, will be assessed by the proportion of monthly urine samples negative vs. positive/missing

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Springer, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale School of Medicine, New Haven, Connecticut
  - UT Southwestern, Dallas, Texas
  - Texas Christian University, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Villaire S, Sease T, Pankow J, Bennett A, Pulitzer Z, Hansen L, Frank C, Di Paola A, Lehman W, Sanchez M, McQuaid A, Schultheis A, Stein B, Springer SA, Nijhawan AE, Knight K. A qualitative examination of barriers and facilitators to HIV prevention and treatment for people involved with the criminal justice system. Health Justice. 2025 Jun 6;13(1):37. doi: 10.1186/s40352-025-00344-6. PMID 40478391
- [Derived] Springer SA, Nijhawan AE, Knight K, Kuo I, Di Paola A, Schlossberg E, Frank CA, Sanchez M, Pankow J, Proffitt RP, Lehman W, Pulitzer Z, Thompson K, Violette S, Harding KK; ACTION Cooperative Group. Study protocol of a randomized controlled trial comparing two linkage models for HIV prevention and treatment in justice-involved persons. BMC Infect Dis. 2022 Apr 15;22(1):380. doi: 10.1186/s12879-022-07354-x. PMID 35428213